CLINICAL TRIAL: NCT06638372
Title: Caffeinated Chewing Gum on Special Forces Performance: a Cross-over Study
Brief Title: Caffeinated Chewing Gum on Special Forces Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Responsible Party: Principal Investigator, Chih-Hui Chiu, Professor, National Taiwan Sport University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 113-7
Record Dates: First submitted 2024-10-05; First posted 2024-10-15 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Caffeine; Placebo
Keywords: exercise performance
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- caffeine gum (Experimental): Chewing caffeine gum for 10 minutes
  Interventions: Dietary Supplement: caffeine
- placebo gum (Placebo Comparator): Chewing placebo gum for 10 minutes
  Interventions: Dietary Supplement: caffeine

INTERVENTIONS:
Dietary Supplement: caffeine — The participants chewing either caffeine Gum (CAF trial, containing 3 mg/kg of caffeine) or Placebo Gum (PL) for 10 minutes. After rested for 15 minutes, the participants underwent tests.

SUMMARY:
The purpose of this project is to investigate the effects of caffeine chewing gum on the cognitive functions and special operations capabilities of special forces.

DETAILED DESCRIPTION:
Using a randomisation crossover design, 20-40 active-duty special forces members who had undergone leave and special forces reserve training were divided into a caffeine trial (CAF) and a placebo trail (PL). After chewing caffeine-containing gum containing 5 mg/kg (CAF group) or caffeine-free gum (PL group) for 15 minutes, then performed a simple reaction test, a stroop test, a visual search test, a grip strength test, a vertical jump test, a 20-metre sprint test, and a counter-terrorism simulation test. A heart rate monitor was used to measure the heart rate and heart rate variability of the participants. Saliva samples were collected and analysed for α-Amylase, cortisol and caffeine concentrations before the test, after a 15-minute break from chewing gum and at the end of the test. Completion time of cognitive functions, grip strength, vertical jump height, 20 m sprint time, time to completion of the counterterrorism simulation test, and target score will be analysed using paired-sample t-tests.

ELIGIBILITY:
Inclusion Criteria:

* Active Special Warfare Unit members who have passed the Grade A Special Forces Reserve Training
* No cardiovascular and joint diseases
* Adult male over 20 years old

Exclusion Criteria:

* Non-active Special Warfare Unit members
* Have cardiovascular and joint diseases
* Under age

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male subjects
Enrollment: 16 (Actual)
Dates: Start 2024-10-05 (Actual); Primary Completion 2024-10-06 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Stroop task | 15 minutes after intervention
  The color-word Stroop task were conducted using Psych/Lab for Windows. The reaction time (millisecond) were recorded.
visual search test | 15 minutes after intervention
  The visual search test were conducted using Psych/Lab for Windows. The reaction time (millisecond) were recorded.

SECONDARY OUTCOMES:
anti-terrorist operations | 15 minutes after intervention
  Target shooting and target finding. The completed time (seconds) were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: ChihHui Chiu, PhD, Principal Investigator — Professor
Locations (1):
- National Taiwan University of Sport, Taichung, North, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-10-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT06638372/Prot_000.pdf